CLINICAL TRIAL: NCT02274012
Title: Phase II Trial of Afatinib in Combination With Weekly Paclitaxel in the Second Line Treatment of HER2 Amplified Advanced Gastric, Gastroesophageal Junction and Esophageal Cancer
Brief Title: Trial of Afatinib in Combination With Weekly Paclitaxel in the Second Line Treatment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Former PI left institution and had plans to continue at another institution.
Sponsor: Columbia University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Naiyer Rizvi, Assistant Professor, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAM5905; 1200.203 (Other: Boehringer Ingelheim Pharmaceuticals, Inc.)
Record Dates: First submitted 2014-10-15; First posted 2014-10-24 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: HER-2 Positive Gastric Cancer; Gastrooesophageal Cancer; Esophageal Cancer
Keywords: Gastric; Gastroesophageal Junction; Gastroesophageal Cancer; Esophageal Cancer; Metastatic; HER2 amplified; Afatinib
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasm Metastasis | interventions — Afatinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Afatinib and weekly Paclitaxel (Experimental): In addition to the standard chemotherapy, afatinib 40 mg orally once daily will be administered starting on the first day of paclitaxel. Translational studies to assess circulating tumor cells at the start of therapy and then at several later time points, including at the time of progression. These studies will assess the correlation of circulating tumor cell numbers with radiographic response and pilot studies will also be conducted to assess HER2 expression, HER2 genomic amplification, HER2 pathway activation and secondary genetic changes in the HER2 coding sequence as well as other pathway components.
  Interventions: Drug: Afatinib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Afatinib — Afatinib 40mg/PO daily will be administered in combination to standard of care paclitaxel.
  Other Names: BIBW 2992
Drug: Paclitaxel — On the day of the first dose of afatinib, paclitaxel will be administered at a dose of 80 mg/m2 intravenously over 60 minutes on days 1, 8 and 15 of a 28-day cycle.
  Other Names: Taxol

SUMMARY:
The investigators are doing this research program to find out if the investigational drug, afatinib which is a medication known to block the function of the ErbB2 protein might help standard chemotherapy, in particular paclitaxel, work better.

Afatinib (GILOTRIF) is a highly potent, irreversible inhibitor of the EGFR and HER2. On July 12, 2013 the United States Food and Drug Administration (US FDA) approved afatinib for the first-line treatment of patients with metastatic non-small cell lung cancer whose tumors had specific EGFR gene mutations (exon 19 deletions or exon 21 i.e. L858R substitution mutations) as detected by an FDA approved test.

Paclitaxel is a standard, anti-cancer medicine that has been approved by the US Food and Drug Administration (FDA) for the treatment of lung cancer.

The combination of Afatinib and Paclitaxel are considered investigational when used in this research program. An investigational drug is a drug that is not approved by the FDA for its indication.

DETAILED DESCRIPTION:
Standard Procedures:

Subjects are offered second line chemotherapy with paclitaxel 80 mg/m2 intravenous infusion over 60 minutes on days 1, 8, and 15 of a 28-day cycle until disease progression or intolerable toxicity.

Experimental Procedures:

In addition to the standard chemotherapy, afatinib 40 mg orally once daily will be administered starting on the first day of paclitaxel. Translational studies to assess circulating tumor cells at the start of therapy and then at several later time points, including at the time of progression. These studies will assess the correlation of circulating tumor cell numbers with radiographic response and pilot studies will also be conducted to assess HER2 expression, HER2 genomic amplification, HER2 pathway activation and secondary genetic changes in the HER2 coding sequence as well as other pathway components.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma or poorly differentiated carcinoma of the intrathoracic esophagus, gastrointestinal junction or stomach.
* Tumor must be HER2 positive 3+ by immunohistochemistry or positive by Fluorescence in situ hybridization (FISH) analysis if 2+ by immunohistochemistry.
* Received and failed at least one prior cytotoxic chemotherapy regimen for advanced disease that included trastuzumab.
* Age greater than or equal to 18 years.
* At least one measurable lesion as defined by modified RECIST criteria.
* ECOG performance status less than or equal to 2.
* Life expectancy of at least 12 weeks.
* Normal organ and marrow function as defined.
* Able to swallow and retain oral medication.
* Left ventricular ejection fraction (LVEF) within institutional range of normal as measured by echocardiogram (ECHO).
* Prior malignancy is acceptable if the subject is considered to be cured.
* Ability to understand and the willingness to sign a written informed consent document.
* All subjects of childbearing potential must agree to use acceptable methods of birth control (Men and Women).
* Willingness to consent to the use of baseline diagnostic tumor specimen for correlative studies.

Exclusion Criteria:

* Squamous cell carcinoma.
* History of clinically relevant cardiovascular abnormalities within 6 months.
* Baseline (less than 1 month before treatment) cardiac left ventricular function with resting ejection fraction of less than 50 percent measured by multigated blood pool imaging of the heart (MUGA scan) or echocardiogram.
* Pregnant and lactating women are excluded from the study.
* Significant or recent acute gastrointestinal disorders with diarrhea.
* More than 2 prior cytotoxic chemotherapy regimens for relapsed or metastatic disease.
* Major surgery, chemotherapy, radiation therapy or other cancer therapy within 3 weeks of treatment day 1.
* Use of any investigational drug within 4 weeks.
* Prior treatment with taxanes if given as full-dose chemotherapy for advanced disease.
* Prior treatment with afatinib or any other HER2 inhibitor other than trastuzumab.
* Front-line chemotherapy that did not contain trastuzumab.
* Active central nervous system disease (CNS) metastases.
* Planned concurrent anti-cancer therapy while taking investigational treatment.
* Unresolved or unstable, serious toxicity from prior cancer treatment (any toxicities greater than grade 2).
* Peripheral neuropathy of Grade 2 or greater
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety.
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to paclitaxel
* Prior anthracycline therapy with a cumulative dose of doxorubicin (or equivalent) greater than or equal to 400 mg/m2
* Pre-existing or current interstitial lung disease
* Known Hypersensitivity to Afatinib (BIBW 2992) or the excipients of any of the trial drugs.
* Patients unable to comply with the protocol.
* Active hepatitis B infection, active hepatitis C infection or known human immunodeficiency virus HIV carrier.
* Known or suspected active drug or alcohol abuse.
* Concomitant treatment with strong inhibitors or inducers of P-glycoprotein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05-29 (Estimated); Primary Completion 2015-08-12 (Actual); Study Completion 2015-08-12 (Actual)

PRIMARY OUTCOMES:
Change of tumor burden (in centimeters) for participants during protocol therapy | Change from Baseline Tumor burden, measured every 8 weeks, up to approximately 4 years

SECONDARY OUTCOMES:
Number of participants with adverse events. | up to approximately 36 months
  Safety of BIBW 2992 will be evaluated as indicated by intensity and incidence of adverse events, graded according to US National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) Version 4.0. Safety endpoints include:
  * events leading to dose reduction
  * events leading to permanent treatment discontinuation
  * the overall incidence and CTC criteria grade of adverse events, as well as relatedness of adverse events to treatment
  * causes of death
Total number of circulating tumor cell (CTC) numbers. | up to approximately 36 months
  CTC number changes from cycle 1, day 1 to cycle 2/3, day 1 will be correlated with response rate, progression-free survival as well as skin toxicity.
Clinical benefit in progression free survival. | every 3 months up to approximately 4 years
Clinical benefit in overall survival. | every 3 months up to approximately 4 years
ErbB2 levels benefit during therapy. | up to approximately 4 years
  Diagnostic tumor specimens will be retrieved for all subjects participating in the protocol. These specimens will be used for confirmation of ErbB2 status as well as correlative analyses of clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Naiyer Rizvi, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Herbert Irving Comprehensive Cancer Center (HICCC) Clinical Trials Page — http://www.hiccc.columbia.edu/clinical-trials